CLINICAL TRIAL: NCT01863979
Title: New Causes and Predictors for the Development of Atrial Fibrillation and Its Complications
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: RMB-0514-12
Record Dates: First submitted 2013-05-12; First posted 2013-05-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Complications of Atrial Fibrillation
Keywords: Atrial Fibrillation; Thromboembolism
MeSH Terms: conditions — Atrial Fibrillation; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Atrial Fibrillation

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia and its prevalence increases with aging of the population. It is reflected in the ECG recording by the replacement of regular P-waves by an undulating baseline and irregular ventricular complexes [2]. The uncoordinated atrial activity prevents effective atrial contraction, leading to clot formation. Atrial fibrillation contributes significantly to population morbidity and mortality, and presently available therapeutic approaches have major limitations, including limited efficacy and potentially serious side effects. It can be classified into one of the three following categories:

1. Paroxysmal: self-termination within 7 days
2. Persistent: requires termination by pharmacological or direct-current electric cardioversion
3. Permanent: restoration to sinus rhythm is impossible or inadvisable

It is believed that in many cases the natural history of AF involves evolution from paroxysmal to persistent to permanent forms through the influence of atrial remodeling caused by the arrhythmia itself and/or progression of underlying heart disease. As many underlying conditions contribute to the development and progression of AF, the full and exact mechanisms standing behind this common arrhythmia are not completely or sufficiently understood.

Thromboembolism is by far the most important complication of AF, and the most common factor in stroke in the elderly. The determinants of Virchow triad, including stasis, endothelial damage, and coagulation properties, are centrally involved in AF- related thrombus formation.

Hence, thorough searching for new possible causes or contributing factors for the developing and progression of AF and its most threatening complication, thromboembolism, is mandatory

The aim of the study is to look for new possible causes of atrial fibrillation and its complications.

DETAILED DESCRIPTION:
This is an observational historical prospective study. All patients admitted to the Rambam health care campus between 1.1.2007 and 31.11.2011 with the primary diagnosis with Acute Atrial Fibrillation and were 18 years old or older at the time of diagnosis, will be included in this historical prospective study.

Patients' demographic data, medical history, permanent medications, laboratory studies, electrocardiographic and echocardiographic reports will be collected from the radiologic information system; a computed medical registry.

After collecting the data, statistical analysis will be performed aiming to discover possible causes or predictors for atrial fibrillation development and the occurrence of its adverse complications, especially thromboembolism.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis with Acute Atrial Fibrillation
* 18 years old or older at the time of diagnosis
* admitted between 1.1.2007 and 31.12.2011

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the Rambam health care campus between 1.1.2007 and 31.12.2011 with the primary diagnosis with Acute Atrial Fibrillation and were 18 years old or older at the time of diagnosis, will be included in this historical prospective study
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Readmission due to Atrial Fibrillation | 3 years

SECONDARY OUTCOMES:
Developement of stroke or transient ischemic attack, Developement of Congestive heart failure and Death | 3 years

REFERENCES:
- [Background] Miyasaka Y, Barnes ME, Gersh BJ, Cha SS, Bailey KR, Abhayaratna WP, Seward JB, Tsang TS. Secular trends in incidence of atrial fibrillation in Olmsted County, Minnesota, 1980 to 2000, and implications on the projections for future prevalence. Circulation. 2006 Jul 11;114(2):119-25. doi: 10.1161/CIRCULATIONAHA.105.595140. Epub 2006 Jul 3. PMID 16818816
- [Background] Wakili R, Voigt N, Kaab S, Dobrev D, Nattel S. Recent advances in the molecular pathophysiology of atrial fibrillation. J Clin Invest. 2011 Aug;121(8):2955-68. doi: 10.1172/JCI46315. Epub 2011 Aug 1. PMID 21804195
- [Background] Dobrev D, Nattel S. New antiarrhythmic drugs for treatment of atrial fibrillation. Lancet. 2010 Apr 3;375(9721):1212-23. doi: 10.1016/S0140-6736(10)60096-7. Epub 2010 Mar 22. PMID 20334907
- [Background] Nattel S, Burstein B, Dobrev D. Atrial remodeling and atrial fibrillation: mechanisms and implications. Circ Arrhythm Electrophysiol. 2008 Apr;1(1):62-73. doi: 10.1161/CIRCEP.107.754564. No abstract available. PMID 19808395
- [Background] de Vos CB, Pisters R, Nieuwlaat R, Prins MH, Tieleman RG, Coelen RJ, van den Heijkant AC, Allessie MA, Crijns HJ. Progression from paroxysmal to persistent atrial fibrillation clinical correlates and prognosis. J Am Coll Cardiol. 2010 Feb 23;55(8):725-31. doi: 10.1016/j.jacc.2009.11.040. PMID 20170808
- [Background] Nattel S, Opie LH. Controversies in atrial fibrillation. Lancet. 2006 Jan 21;367(9506):262-72. doi: 10.1016/S0140-6736(06)68037-9. PMID 16427496
- [Background] Watson T, Shantsila E, Lip GY. Mechanisms of thrombogenesis in atrial fibrillation: Virchow's triad revisited. Lancet. 2009 Jan 10;373(9658):155-66. doi: 10.1016/S0140-6736(09)60040-4. PMID 19135613